CLINICAL TRIAL: NCT00950235
Title: Weight Management for Improved Pregnancy Outcomes
Acronym: Healthy Moms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01HD058061-01A1 (NIH); 1R01HD058061 (NIH)
Record Dates: First submitted 2009-07-29; First posted 2009-07-31 (Estimated); Results first posted 2015-07-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-06

CONDITIONS: Obesity; Pregnancy
Keywords: obese; pregnant; large for gestational age; large for gestational age baby
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Other): This arm will receive one additional nutrition counseling session that typically received in the health system. This arm will be compared to our intervention group
  Interventions: Other: Usual Care
- Weight Management Counseling (Experimental): In-person and group session counseling
  Interventions: Behavioral: Weight Management

INTERVENTIONS:
Behavioral: Weight Management — Two individual counseling session on nutrition and once weekly group sessions including use of food diaries for the remaining weeks of their pregnancy
  Arms: Weight Management Counseling
Other: Usual Care — Standard nutrition counseling from Health Plan
  Arms: Usual Care

SUMMARY:
This study will examine the safety and effectiveness of a dietary intervention in pregnant women. Women who are obese will be invited to participate. The control arm will receive routine prenatal care and one in-person nutritional and dietary counseling session to promote healthy eating during their pregnancy. The intervention arm will receive a more intensive dietary program that will include in-person counseling and group support sessions. The goal of the intervention will be weight maintenance (weight at 2 weeks after delivery should be within 3% of baseline weight) and avoidance of postpartum weight retention

ELIGIBILITY:
Inclusion Criteria:

* BMI 30 or more
* Less than 20 weeks gestation
* member of Kaiser Permanente Northwest (NW)
* receive pre-natal care at Kaiser Permanente NW
* speaks English

Exclusion Criteria:

* no current treatment for cancer
* no bariatric surgery
* no current renal disease
* no multiple birth anticipated
* no hyperemesis requiring hospitalization
* no diabetes (type 1 or 2)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2009-10; Primary Completion 2012-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor J Stevens, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States

REFERENCES:
- [Derived] Vesco KK, Karanja N, King JC, Gillman MW, Leo MC, Perrin N, McEvoy CT, Eckhardt CL, Smith KS, Stevens VJ. Efficacy of a group-based dietary intervention for limiting gestational weight gain among obese women: a randomized trial. Obesity (Silver Spring). 2014 Sep;22(9):1989-96. doi: 10.1002/oby.20831. PMID 25164259
- [Derived] Vesco KK, Karanja N, King JC, Gillman MW, Perrin N, McEvoy C, Eckhardt C, Smith KS, Stevens VJ. Healthy Moms, a randomized trial to promote and evaluate weight maintenance among obese pregnant women: study design and rationale. Contemp Clin Trials. 2012 Jul;33(4):777-85. doi: 10.1016/j.cct.2012.03.006. Epub 2012 Mar 20. PMID 22465256

RESULTS

PARTICIPANT FLOW:
Recruitment Details: English speaking, obese, age 18 or older receiving pregnancy care at an prepaid health plan clinic. Less than 21 weeks gestation. Recruitment November 2009-July 2011.
Pre-assignment Details: Women were invited to attend an informational meeting which explained the study and covered the elements of consent. Interested volunteers were asked to come back to the research setting for the baseline visit. Randomization occurred at the baseline visit after a final review of eligibility and signing a consent.
Period: Overall Study
Arm/Group | Usual Care | Weight Management Counseling
Started | 60 | 58
Completed | 58 | 54
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Weight Management Counseling | Total
Number analyzed (Participants) | 60 | 58 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 58 | 118
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 58 | 118
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 53 | 52 | 105
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 51 | 50 | 101
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 60 | 58 | 118
Weight [Mean (Standard Deviation); unit: kg] | 100.5 (15.6) | 98.8 (15.1) | 99.7 (15.3)

OUTCOME MEASURES:

1. Primary Outcome: Maternal Weight Change
Description: We chose the weight at 2 weeks postpartum, rather than at an end point during pregnancy, to avoid the contribution of products of conception, maternal edema, and increased maternal blood volume to the weight gain.
Time Frame: baseline to 2 weeks post partum
Population: Data was from follow up visit or validated clinical data
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care | Weight Management Counseling
Number analyzed (Participants) | 58 | 56
kg | 1.2 (5.6) | -2.6 (5.5)

2. Secondary Outcome: Pregnancy Weight Change
Time Frame: baseline to 34 weeks gestation
Population: Participants returning for follow up visit or validated clinical data
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care | Weight Management Counseling
Number analyzed (Participants) | 58 | 56
kg | 8.4 (4.7) | 5.0 (4.1)

3. Secondary Outcome: Large for Gestational Age (LGA)
Description: Large-for-gestational-age defined as weight greater than the 90th percentile for gestational age at birth.
Time Frame: At birth
Population: Babies born to participants
Measure: Number; unit: participants
Arm/Group | Usual Care | Weight Management Counseling
Number analyzed (Participants) | 58 | 56
participants | 15 | 5

ADVERSE EVENTS:
Time Frame: AE data collected at follow up visits (34wk gestation, 2 weeks post-partum, 6 and 12 months post partum)
Description: AE data collected between November 2009 and July 2011, 20 months
Arm/Group | Usual Care | Weight Management Counseling
Serious Adverse Events (participants affected / at risk) | 2/60 | 0/58
Other Adverse Events (participants affected / at risk) | 40/60 | 30/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=60) | Weight Management Counseling (N=58)
miscarriage (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=60) | Weight Management Counseling (N=58)
Cesarean Section (Pregnancy, puerperium and perinatal conditions) | 26 (26) | 21 (21)
Pre-Term Birth <37 weeks (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 4 (4)
NICU admission (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 2 (2)
Respiratory morbidity (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No